CLINICAL TRIAL: NCT03848780
Title: Pharmacological Preconditioning With Desflurane in Liver Surgery
Brief Title: Desflurane Preconditioning in Hepatectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Eleni Koraki, Principal investigator, Anesthesiologist, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 3779
Record Dates: First submitted 2019-01-29; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Ischemia Reperfusion Injury
Keywords: preconditioning; hepatectomy; ischemia reperfusion injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Desflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane Group (Experimental): Thirty minutes before initiation of ischemia the surgeon was instructed to notify the anesthesiologist. At this single time point, propofol infusion was stopped and substituted with the volatile anesthetic desflurane to achieve a Minimum Alveolar Concentration of 1. The procedure included a 5-minute induction of desflurane, a 20-minute preconditioning and a 5-minute washout period when propofol was reintroduced and desflurane stopped.
  Interventions: Drug: Desflurane
- Control Group (No Intervention): No pharmacological preconditioning was implemented

INTERVENTIONS:
Drug: Desflurane
  Arms: Desflurane Group

SUMMARY:
Hepatectomies are considered as operations of high bleeding risk. The history of massive hemorrhage in liver surgery led to the emergence of techniques to control excessive blood loss. These techniques temporarily occlude the blood vessels that supply liver (the Pringle Maneuver) limiting subsequent losses. However, this leads to the ischemia - reperfusion injury impairing liver function. Research points to methods targeting on tempering reperfusion pathophysiology. Volatile anesthetics have been used for pharmacological preconditioning and proved to protect against organ damage. The aim of this study was to investigate the potential beneficial effect of desflurane on ischemia-reperfusion injury of the liver. Patients presenting for elective hepatectomy were randomized equally into two groups. The Control Group received no pharmacological preconditioning and the Desflurane Group received pharmacological preconditioning with Desflurane before induction of ischemia.

DETAILED DESCRIPTION:
Hepatectomies are characterized by an elevated risk of severe hemorrhage. The high vascular supply of the liver has historically troubled surgeons who resolved to techniques to control excessive blood loss. The Pringle Maneuver commonly employed in liver surgery is a temporary method to occlude the vascular supply of the liver. As a result, ischemia is developed and a pathophysiologic cascade is initiated. Upon the resolution of ischemia, reperfusion occurs which is linked to further damage and the ischemia-reperfusion injury is developed. Ischemia and reperfusion lead to activation of the innate immune response, which interacts with the adaptive immune response. Result of this interaction is the production of inflammatory cytokines, chemokines, complement products, and the recruitment of neutrophils to the site of injury. Previous studies have shown that animal's livers suffered from ischemia-reperfusion injury had increased neutrophil infiltration and pharmacological agents attenuating neutrophil's activity improved hepatic Ischemia-Reperfusion Injury (IRI). Preconditioning refers to the exposure of an organ to short intervals of ischemia which has been shown to mitigate the aforementioned ischemia-reperfusion injury. Preconditioning can be pharmacological and volatile anesthetics have been successfully used in preconditioning models. Sevoflurane have been proved beneficial for a series of hepatectomies in limiting transaminase levels postoperatively. However, sevoflurane by virtue can be hepatotoxic through Compound A production, elevated free calcium and reactive oxide species activation. On the other hand, desflurane undergoes minimum liver metabolism. In liver ischemia-reperfusion models, desflurane preconditioning led to decreased cell death and inflammatory cytokines inhibition.

The goal of the investigator's study was to investigate the effect of desflurane preconditioning in patients undergoing elective hepatectomy of at least two segments. Patients were randomized 1:1 to receive pharmacological preconditioning (Desflurane Group, Group D) or not (Control Group, Group C). The surgeon and the Intensive Care Unit were blinded as to the intervention. Anesthetic management was the same for all patients. For GroupD thirty minutes before the initiation of ischemia desflurane was delivered and propofol was stopped for the same interval.

ELIGIBILITY:
Inclusion Criteria:

* hepatectomy of at least two segments

Exclusion Criteria:

* Hepatitis B, C or HIV infection
* liver cirrhosis
* autoimmune disease, inflammatory bowel disease
* pregnancy
* prior additional ablation therapies (cryosurgery or radiofrequency)
* liver resections without inflow occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Matrix Metalloproteinases (MMPs) 2 and 9 level | Sample 1: At surgery, before initiation of the procedure , Sample 2: Thirty minutes after reperfusion
  The levels of Matrix Metalloproteinase 2 and Matrix Metalloproteinase 9 as evaluated by the relative gene expression using RT-PCR. The comparative CT method also referred to as the 2-ΔΔCT method was used to calculate the fold change and then convert it to percentage. Their presence has been linked to hepatic cellular injury so increased levels represent worse injury.
Tissue Inhibitor Metalloproteinase (TIMPs) 1and 2 | Sample 1: At surgery, before initiation of the procedure , Sample 2: Thirty minutes after reperfusion
  The levels of Tissue Inhibitor Metalloproteinase 1 and Tissue Inhibitor Metalloproteinase 2 as evaluated by the relative gene expression using RT-PCR. The comparative CT method also referred to as the 2-ΔΔCT method was used to calculate the fold change and then convert it to percentage. Their inhibitory effect on Matrix Metalloproteinases has been associated with a limitation of cellular injury. Thus, the higher the levels of Tissue Inhibitor Metalloproteinases the greater their protective activity.

SECONDARY OUTCOMES:
Histological findings of hepatic parenchyma | Sample 1: Upon surgical dissection of the liver, before inflow occlusion, Sample: thirty minutes after reperfusion
  Hematoxylin Eosin, Gomori and Μasson staining were used. With Hematoxylin Eosin staining the degree of steatosis was assessed while Gomori and Masson staining was used to determine the level of fibrosis.
  Steatosis was characterized (x100 magnification) as mild (10%-30%), moderate (30%-60%), severe (>60%) according to the presence of fat droplets in hepatic cells.
  Fibrosis was also graded based on the METAVIR score as absent - F0, portal fibrosis without septa - F1, portal fibrosis with rare septa - F2, numerous septa - F3 and cirrhosis - F4.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Koraki, Dr, Principal Investigator — Aristotle University Of Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen HR, Martin P, Goss J, Donovan J, Melinek J, Rudich S, Imagawa DK, Kinkhabwala M, Seu P, Busuttil RW, Shackleton CR. Significance of early aminotransferase elevation after liver transplantation. Transplantation. 1998 Jan 15;65(1):68-72. doi: 10.1097/00007890-199801150-00013. PMID 9448146
- [Background] Kimura F, Shimizu H, Yoshidome H, Ohtsuka M, Kato A, Yoshitomi H, Nozawa S, Furukawa K, Mitsuhashi N, Sawada S, Takeuchi D, Ambiru S, Miyazaki M. Circulating cytokines, chemokines, and stress hormones are increased in patients with organ dysfunction following liver resection. J Surg Res. 2006 Jun 15;133(2):102-12. doi: 10.1016/j.jss.2005.10.025. Epub 2006 Jan 4. PMID 16386757
- [Background] Boros P, Bromberg JS. New cellular and molecular immune pathways in ischemia/reperfusion injury. Am J Transplant. 2006 Apr;6(4):652-8. doi: 10.1111/j.1600-6143.2005.01228.x. PMID 16539620
- [Background] Beck-Schimmer B, Breitenstein S, Urech S, De Conno E, Wittlinger M, Puhan M, Jochum W, Spahn DR, Graf R, Clavien PA. A randomized controlled trial on pharmacological preconditioning in liver surgery using a volatile anesthetic. Ann Surg. 2008 Dec;248(6):909-18. doi: 10.1097/SLA.0b013e31818f3dda. PMID 19092335

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT03848780/Prot_SAP_000.pdf